CLINICAL TRIAL: NCT05963217
Title: Phase I/Ib Study of TBI-2001 for Patients With Relapsed or Refractory CD19+ B-cell Lymphoma, Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL)
Brief Title: Study of TBI-2001(Autologous CD19 Specific Chimeric Antigen Receptor (CAR) Gene-transduced T Lymphocytes) for Relapsed or Refractory CD19+ B-cell Lymphoma, CLL/SLL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBI-200101
Record Dates: First submitted 2023-06-27; First posted 2023-07-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Relapsed or Refractory CD19+ B-cell Lymphoma; Relapsed or Refractory Chronic Lymphocytic Leukemia; Relapsed or Refractory Small Lymphocytic Lymphoma
Keywords: CD19+ B-cell Lymphoma; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL; Lymphoma; TBI-2001; Anti-CD19 CAR Expressing T cell Therapy; CD19 CAR Gene-Transduced Lymphocyte; Adoptive Immunotherapy; Genetically Engineered Lymphocyte Therapy; Retroviral Vector; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Experimental; Immune System Diseases; Chimeric Antigen Receptor
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Experimental; Immune System Diseases | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Dose Level 1 to 3 (Experimental): 0.3 to 3 x 10^6 autologous CD19-CAR-T cells/kg per patient will be administered intravenously after a conditioning chemotherapy with cyclophosphamide and fludarabine.
  Interventions: Biological: TBI-2001; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: TBI-2001 — Phase-I portion:
  cohort 1: 3×10^5 cells/kg, cohort 2: 1×10^6 cells/kg, cohort 3: 3×10^6 cells/kg). Phase-Ib portion: The dose of Phase-Ib will be determined during the phase I portion.
Drug: Cyclophosphamide — IV Cyclophosphamide (for 3 days) will be administered as conditioning before cell infusion with TBI-2001.
Drug: Fludarabine — IV Fludarabine (for 3 days) will be administered as conditioning before cell infusion with TBI-2001.

SUMMARY:
This is a Phase 1/1b, open-label, dose-escalation study to evaluate the safety and the efficacy of anti-CD19 chimeric antigen receptor (CAR) (TBI-2001) for relapsed or refractory CD19+ B-cell lymphoma Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL).

DETAILED DESCRIPTION:
TBI-2001 is a next-generation CAR-T product including costimulatory sequences that lead to the activation of cytokine-related JAK/STAT signaling pathways. This is a first-in-human study of TBI-2001 and will follow a 3+3 design of dose-escalation cohorts. Additional subjects will be treated with TBI-2001 at the determined recommended phase 2 dose (RP2D) following cyclophosphamide and fludarabine pre-treatment. Long-term follow-up is conducted for 5 years following the infusion of TBI-2001

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed CD19 positive B cell Non-Hodgkin Lymphoma (NHL), Chronic Lymphocytic Leukemia (CLL), or Small Lymphocytic Lymphoma (SLL) who have received at least 2 prior therapies.
2. Phase Ib cohort will enroll CLL/SLL patients only.
3. ECOG Performance Status 0 or 1.
4. Age ≥18 years at time of consent.
5. Life expectancy greater than 4 months.
6. For cessation of therapies prior to apheresis and lymphodepleting chemotherapy (bridging therapies), the institutional (UHN) SOPs related to Kymriah will be followed. However, an exception will be made for targeted and biological therapies that decrease circulating disease and are not expected to negatively impact successful harvest of lymphocytes by apheresis. In these cases, after discussion with and approval by the Sponsor, no washout will be required.
7. Patients must have adequate key organ function (bone marrow, heart, lung, liver, renal, etc)
8. Consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
9. The treating investigator should consider the patient to have disease that is incurable, and that the patient would be a reasonable candidate for future treatment with TBI-2001 within the next 3 months

Exclusion Criteria:

1. Uncontrolled intercurrent illnesses or medical conditions that may interfere with trial participation.
2. Active or prior documented autoimmune disease within the past 2 years.
3. History of primary immunodeficiency.
4. History of organ transplant that requires use of immunosuppressive medications.
5. History hypersensitivity to components of manufacture or excipients of investigational drug.
6. Untreated central nervous system (CNS) metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids.
7. Other invasive malignancy within 2 years except for noninvasive malignancies
8. Current or prior use of immunosuppressive medication within 14 days before apheresis.
9. Any condition that, in the opinion of the investigator, would interfere with the evaluation of TBI-2001 or interpretation of subject safety or study results.
10. Known history of untreated active tuberculosis.
11. HIV positivity.
12. Active HTLV or syphilis infection.
13. Active hepatitis B or active hepatitis C. Subjects with a negative PCR assay for viral load for hepatitis B or C are permitted.
14. Pregnant or lactating women.
15. Received allogeneic-HSCT.
16. Any prior CD19 directed therapy.
17. Live vaccine within 28 days prior to apheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety of TBI-2001 | One month
  Dose Limiting Toxicities (DLTs)
Safety of TBI-2001 | One year
  Adverse event (AEs)
Safety of TBI-2001 | One year
  Laboratory testing- RCR appearance and Clonality
Recommended phase 2 dose (RP2D) of TBI-2001 | One year
  RP2D to be determined during the dose escalation cohort

SECONDARY OUTCOMES:
Efficacy of TBI-2001; Overall Response Rate (ORR) | One year
  Overall Response Rate (ORR) (Complete Response (CR)+Partial Response(PR))
Efficacy of TBI-2001; Durable Response Rate (DRR) | One year
  Durable Response Rate (DRR) as defined as CR or PR sustained for at least 6 months
Efficacy of TBI-2001; Progression free survival (PFS) | One year
  Progression free survival
Efficacy of TBI-2001; Overall survival (OS) | One year
  Overall survival

OTHER OUTCOMES:
Persistence of TBI-2001 | One year
  Percentage of CAR T in peripheral blood and bone marrow using PCR and Flow cytometry.
Minimal residual disease (MRD) negative rate (in CLL patients) | One year
  MRD negative rate

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Butler, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No